CLINICAL TRIAL: NCT05322395
Title: Safety and Feasibility of Triage and Rapid Discharge of Patients With Chest Pain From Accident and Emergency: a Pragmatic, Randomised, Multicentre, Non-inferiority Control Trial of the Accelerated European Society of Cardiology (ESC) 0-1 Hour Pathway vs. Conventional 0-3 Hour Accelerated Diagnostic Protocol.
Brief Title: Pragmatic Randomised Trial of the ESC 0/1 Versus 0/3 Hour Troponin Pathway
Acronym: MACROS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: northwest coast academic science network (Unknown); Quidel Corporation (Industry); Siemens Corporation, Corporate Technology (Industry); Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPO635
Record Dates: First submitted 2022-01-04; First posted 2022-04-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Acute Coronary Syndrome; Troponin; Chest Pain; Point-of-care Systems
Keywords: acs; POC troponin; high sensitivity troponin
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Intervention Model Description: A two-arm parallel group, two-centre randomised controlled trial of 0-1-hour high sensitivity troponin T (hs cTnT) compared to a 0-3-hour pathway as rules for rapid discharge of suspected ACS. (both incorporating single presentation sample limit of detection (LOD) high sensitive troponin as a rule for discharge, or cut-off selected by manufacturer).
  The power of the study is on safety rather than percent discharge achieved by 4 hours as this is the primary focus for clinicians and health care institutions. (By virtue of the earlier sampling the 0-1 hour troponin sampling is likely to allow greater discharges by 4 hours and the sample size for safety easily accommodates this aspect).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESC 0/1 pathway (Experimental): A two-arm parallel group, two-centre pragmatic randomised controlled trial of 0-1-hour high sensitivity troponin T (hs cTnT) compared to a 0-3-hour pathway as rules for rapid discharge of suspected ACS. (both incorporating single presentation sample limit of detection (LOD) high sensitive troponin as a rule for discharge, or cut-off selected by manufacturer).
  The power of the study is on safety rather than percent discharge achieved by 4 hours as this is the primary focus for clinicians and health care institutions. (By virtue of the earlier sampling the 0-1 hour troponin sampling is likely to allow greater discharges by 4 hours and the sample size for safety easily accommodates this aspect).
  Interventions: Diagnostic Test: ESC 0/1 hour troponin pathway
- ESC 0/3 hour pathway (Active Comparator): A two-arm parallel group, two-centre pragmatic randomised controlled trial of 0-1-hour high sensitivity troponin T (hs cTnT) compared to a 0-3-hour pathway as rules for rapid discharge of suspected ACS. (both incorporating single presentation sample limit of detection (LOD) high sensitive troponin as a rule for discharge, or cut-off selected by manufacturer).
  The power of the study is on safety rather than percent discharge achieved by 4 hours as this is the primary focus for clinicians and health care institutions. (By virtue of the earlier sampling the 0-1 hour troponin sampling is likely to allow greater discharges by 4 hours and the sample size for safety easily accommodates this aspect).
  Interventions: Diagnostic Test: ESC 0/1 hour troponin pathway

INTERVENTIONS:
Diagnostic Test: ESC 0/1 hour troponin pathway — randomisation to 0/1 versus 0/3 hour pathway
  Other Names: esc 0/3 hour troponin pathway

SUMMARY:
The primary objective of this study is to assess the feasibility and impact of implementing the ESC 0-1 hour high sensitive troponin pathway in clinical practice and with specific reference to the 0-3 hour pathway currently in use.

The principal outcome measure will be the safety of the 0-1 hour protocol (which is less established and has limited data on safety when implemented in clinical practice)

DETAILED DESCRIPTION:
1. the investigators propose to compare 2 'gold standard' NICE recommended/ESC guideline-backed pathways; the accelerated 0-1 hour troponin clinical pathway versus the conventional 0-3-hour pathway, in a randomised multicentre controlled study.

   1. The primary outcome is to compare percentage safe (with the emphasis and sample size calculation on safety) discharge by 4 hours from presentation by means of the 0-3 hours versus the 0-1-hour (with the 0 hour in both pathways incorporating discharge using the limit of detection).
   2. the investigators propose to use high sensitivity troponin T (hs cTnT) (ROCHE, Elecsys assay as this is currently in routine clinical use at the site) for this purpose and also perform comparative analyses using a high sensitivity troponin I (hs cTnI) assay (ABBOTT, Architect).
2. Redundant blood sample will also be used to evaluate point of care testing (POCT), with additional blood sample taken for POC. These samples will be undertaken as part of routine clinical care and will not require additional venepuncture (and will only be analysed if consent is gained for tissue use in research) population. A co-primary endpoint will be single sample rule-out by point of care troponin (POCT) (with a value of <4ng/l in those with chest pain onset >3 hours from presentation) as assessed in the recent APACE study of triage true POC.11 A comparison of this rule-out in terms of effectiveness (percentage discharge) and safety (sensitivity) will be made with ROCHE lod (<5ng/l)12 and the optimised rule-out of Abbott architect (HSTNI<5ng/l)13

2.2 Secondary objectives

1. The relative performance of the Abbott Architect high sensitivity troponin I (hs TnI) , Quidel's TriageTrue and Siemens Attellica troponin I assay will also be assessed in terms of the primary and secondary endpoints by reference to high sensitivity troponin T (hs cTnT) with cut-points for Abbott hs-cTn I from the BACC study used for the 0-1-hour pathway.14
2. The performance of the novel machine learning algorithm, the Myocardial Ischemic Injury Index (MI3, Abbott) will also be assessed retrospectively with regard to safety and efficacy. This sub study using fully anonymized data will be performed in association with coinvestigators from Abbott Diagnostics (appendix 1).
3. To understand if low levels of Growth Differentiation Factor (GDF-15), could expand safe discharge beyond the LOD. This will be tested for retrospectively in stored plasma samples.
4. To assess if point of care troponin samples at time points at 1 to 3 hours (additional samples) mirror gold standard high sensitive troponin analysis with respect to diagnosis of acute or chronic myocardial injury and/or type 1 or type 2 myocardial infarction.

3) Hypothesis That an accelerated 0-1-hour troponin protocol, when implemented into clinical practice as a pragmatic RCT, will effect safe discharge with greater numbers discharged, by 4 hours from presentation, compared to the use of the more conventional 0-3 hour troponin protocol.

Means to test hypothesis: A two-arm parallel group, two-centre randomised controlled trial of 0-1-hour high sensitivity troponin T (hs cTnT) compared to a 0-3-hour pathway as rules for rapid discharge of suspected ACS. (both incorporating single presentation sample limit of detection (LOD) high sensitive troponin as a rule for discharge, or cut-off selected by manufacturer).

The power of the study is on safety rather than percent discharge achieved by 4 hours as this is the primary focus for clinicians and health care institutions. (By virtue of the earlier sampling the 0-1 hour troponin sampling is likely to allow greater discharges by 4 hours and the sample size for safety easily accommodates this aspect).

4. Outcomes: 4.1 Primary endpoint

1) the investigators will compare safe discharge by each strategy (ie the ESC 0-1 hour pathway versus 0-3 pathway) and the proportion actually discharged by each pathway at 4 hours. The exact definition of safety will be percentage (of cohort randomised to each pathway) safely discharged by 4 hours of presentation to accident and emergency (Safety will be judged by type 1 myocardial infarction, cardiovascular death by 4 weeks with sensitivity >98% - the study will be powered on safety to establish whether 0-1-hour performance is equivalent to 0-3-hour sampling by means of a non-inferiority analysis- see statistics).

(Type 1 myocardial infarction is due to acute coronary atherothrombotic myocardial injury with either plaque rupture or erosion and, often, associated thrombosis. A separate analysis will also be undertaken with inclusion of type 2 MI as well as type 1 MI as an endpoint

4.2 Co-primary endpoint: There will be a comparison of the real time performance of point of care troponin (POCT) assay to that of a sample sent for analysis in the laboratory (the current gold standard of central laboratory analysis using HS cTn).The primary interest will be in presentation sample POC rule-out (triage true (quidel) POC <4ng/l with CP onset >3 hours compared to LOD or optimised rule-out of ROCHE (elecsys) assay, siemens attelica and Abbott architect. There will be a similar comparison made with siemens VTLI troponin I POC assay using FDA approved cut-points for MI rule-out

4.3 Secondary Endpoints:

1. Type 1 myocardial infarction (adjudicated with the use of Abbott hs cTnI) and cardiovascular death* at 4 weeks (target for safety negative predictive value (NPV) >99.5% and sensitivity >98%). (co-primary endpoint). This analysis will be repeated incorporating both type 1 and 2 MI definition. (prespecified secondary analysis)
2. All cause death, type 1 myocardial infarction and urgent or emergency revascularisation. This analysis will be repeated incorporating both type 1 and 2 MI definition. (prespecified secondary analysis)
3. Proportion with rule-out or rule-in MI in the 0-1 hour and 0-3 hour
4. Prediction of MI with myocardial ischemic injury index (MI3) algorithm9
5. HEART ≤3 and a modified HEART score for rule-out MI at 30 days15
6. Proportion with repeat presentations to accident and emergency within 30 days
7. Proportion undergoing coronary angiography and coronary revascularisation in 0-1 versus 0-3 hour pathway
8. Performance of point of care troponin samples at time points at 1 to 3 hours (additional samples to 0 hour) with respect to diagnosis of acute or chronic myocardial injury and/or type 1 myocardial infarction
9. Rule out of MI with GDF-15 (Growth Differentiation Factor 15)

   * Cardiovascular deaths include deaths that result from an myocardial infarctions (MI), sudden cardiac death, death due to heart failure (HF), death due to stroke, death due to cardiovascular procedures, death due to cardiovascular haemorrhage, and death due to other cardiovascular causes and deaths that do not have a clear non- cardiovascular cause.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain with moderate or high suspicion chest pain (see chest pain evaluation chart at end) or any patient the clinician deems suspicious for myocardial ischaemia thus requesting a troponin sample (between daytime hours 0800hrs to 1800hrs)
* Presentation <12 hours since onset of chest pain (or unknown duration)
* Age >18 years of age

Exclusion Criteria:

* ST elevation myocardial infarction (STEMI) infarct on the presenting electrocardiogram (ECG)
* Symptoms considered definitely non-cardiac
* Trauma
* Pregnancy
* Comorbid conditions requiring hospital admission
* Coronary artery bypass graft surgery (CABG) <1 month
* coexistent clinical conditions likely to preclude follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3536 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
percentage safe discharge by 4 hours. safety defined as type 1 MI and CV deah | 4 hours
  We will compare safe discharge by each strategy (ie the ESC 0-1 hour pathway versus 0-3 pathway) and the proportion actually discharged by each pathway at 4 hours. The exact definition of safety will be percentage (of cohort randomised to each pathway) safely discharged by 4 hours of presentation to accident and emergency (Safety will be judged by type 1 myocardial infarction, cardiovascular death by 4 weeks with sensitivity >98% - the study will be powered on safety to establish whether 0-1-hour performance is equivalent to 0-3-hour sampling by means of a non-inferiority analysis- see statistics).
  (Type 1 myocardial infarction is due to acute coronary atherothrombotic myocardial injury with either plaque rupture or erosion and, often, associated thrombosis. A separate analysis will also be undertaken with inclusion of type 2 MI as well as type 1 MI as an endpoint
point of care troponin performance compared to laboratory performance | 4 hours
  largely rule-out of Quidel triage true and siemens VTLI

SECONDARY OUTCOMES:
Type 1 myocardial infarction | 30 days
All cause death, type 1 myocardial infarction and urgent or emergency revascularisation. This analysis will be repeated incorporating both type 1 and 2 MI definition. (prespecified secondary analysis) | 30 days
Proportion with rule-out or rule-in MI in the 0-1 hour and 0-3 hour | 30 days
Prediction of MI with myocardial ischemic injury index (MI3) algorithm | 30 days
HEART ≤3 and a modified HEART score for rule-out MI at 30 days | 30 days
Proportion with repeat presentations to accident and emergency within 30 days | 30 days
Proportion undergoing coronary angiography and coronary revascularisation in 0-1 versus 0-3 hour pathway | 1 year
Performance of point of care troponin samples at time points at 1 to 3 hours (additional samples to 0 hour) with respect to diagnosis of acute or chronic myocardial injury and/or type 1 myocardial infarction | 30 days
Rule out of MI with GDF-15 (Growth Differentiation Factor 15) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather Rodgers, Study Director — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- liverpool university Hospital nhs foundation trust, Liverpool, GB, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khand A, Hatherley J, Dakshi A, Miller G, Bailey L, Fisher M, Goulden C, Noori Z, Rawat A, Hornby R, Fearon H, Meah N, Davies S, Sekulska K, Hassan A, Lambert A, Phillips S, Raj R, Wiles T, Collinson P. Safety and feasibility of triage and rapid discharge of patients with chest pain from emergency room: A pragmatic, randomized noninferiority control trial of the European Society of Cardiology (ESC) 0 to 1 hour pathway vs conventional 0 to 3 hour accelerated diagnostic protocol. Am Heart J. 2024 Dec;278:235-247. doi: 10.1016/j.ahj.2024.08.005. Epub 2024 Aug 14. PMID 39151715